CLINICAL TRIAL: NCT03231449
Title: A Survey of Hospitalizations in Cardiology Units in Sub-Saharan Africa
Acronym: FEVRIER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cardiologie et Développement (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Xavier Jouven, Professor, Cardiologie et Développement
Other Study IDs: 001
Record Dates: First submitted 2017-07-21; First posted 2017-07-27 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Acute Coronary Syndrome; Heart Failure; Syncope; Stroke; Pericarditis; Endocarditis; Conduction Abnormalities; Rhythm; Abnormal; Pulmonary Embolism; Deep Vein Thrombosis; Other Cardiovascular Conditions
Keywords: routine care, evaluation, Africa, observatory
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure; Syncope; Stroke; Pericarditis; Endocarditis; Arrhythmias, Cardiac; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observation of current care — The study FEVRIER (survey of hospitalizations in cardiology units in sub-Saharan Africa) aims to establish a description of sub-Saharan standard of care, in order to get a cross sectional analysis (globally and per country) and a longitudinal analysis (evolution during 5 years).

SUMMARY:
FEVRIER study is an observatory of hospitalizations in cardiology units in sub-Saharan Africa.

DETAILED DESCRIPTION:
FEVRIER is an observational study based on a questionnaire completed by investigators for each hospitalization in cardiology unit during the month of February.The investigator is a physician of the participating hospital.

FEVRIER evaluates the modalities of care management. It will take place in cardiology units of hospitals of sub-Saharian countries one month per year (month of February) during 5 years.

The investigator will thoroughly complete:

* one information form describing the hospital and the department
* one questionnaire (2o questions) for each hospitalized patient

Patients with at least one day of hospitalization will be enrolled in the study. On the first day of February, all patients already hospitalized will be enrolled and all patients hospitalized in the last day of February will be followed until their discharge. thus, data collection will start 1st day of investigation, during February and will continue until the discharge of the last enrolled patient.

ELIGIBILITY:
Inclusion Criteria:

* to be hospitalized in a cardiology department of a participating center during the month of February

Exclusion Criteria:

* refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Each patient hospitalized in cardiology unit of participating centers during the month of February can be included.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Description of patients in cardiology unit in sub-Saharan Africa:socio-demographic characterization | 5 years
  low/medium low / medium high/high
Description of patients in cardiology unit in sub-Saharan Africa:causes of hospitalization | 5 years
  one answer with main reason for hospitalization
Description of patients in cardiology unit in sub-Saharan Africa: co-morbidities | 5 years
  cardiovascular risk factors/history of cardiovascular disease/kidney disease/cancer/alcoholism/psychiatric disorder/sickle cell anemia/HIV:Hepatitis/tuberculosis/other
Description of patients in cardiology unit in sub-Saharan Africa: hospital examinations | 5 years
  blood test/ECG/Chest Xray/Echocardiography/Coronarography/Brain scan
Description of patients in cardiology unit in sub-Saharan Africa: duration of hospitalization | 5 years
  number of days spent in cardiology departement
Description of patients in cardiology unit in sub-Saharan Africa: discharge diagnosis | 5 years
  medical conclusion

SECONDARY OUTCOMES:
number of patients with heart failure | 5 years
  to measure the evolution of the number of patients with heart failure over 5 years
number of patients with myocardial infarction | 5 years
  to measure the evolution of the number of patients with myocardial infarction over 5 years
number of patients with atrial fibrillation | 5 years
  to measure the evolution of the number of patients with atrial fibrillation over 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Jouven, MD, PhD, Principal Investigator — cardiologie et Developpement
Locations (20):
- Centre national hospitalier et universitaire Koutoukou Maga, Cotonou, Benin
- Centre médical Paul IV, Ouagadougou, Burkina Faso
- Hopital militaire de Kamenge et polyclinique maison médicale, Bujumbura, Burundi
- Cameroon (4):
  - Hôpital Régional, Bafoussam
  - Douala General Hospital, Douala
  - Central Hospital, Yaoundé
  - Hôpital Général de Yaoundé, Yaoundé
- Côte d’Ivoire (2):
  - Institut de Cariologie d'Abidjan, Abidjan
  - CHU, Bouaké
- Democratic Republic of the Congo (2):
  - Clinique Ngaliema, Kinshasa
  - Clinique universitaire de Kinshasa, Kinshasa
- Centre Hospitalier Universitaire (CHUL), Libreville, Gabon
- CHU Ignace Deen, Conakry, Guinea
- Institut du coeur, Maputo, Mozambique
- Hôpital National Lamorde, Niamey, Niger
- CHU, Brazzaville, Republic of the Congo
- Senegal (3):
  - Hôpital de Fann, Dakar
  - Hôpital général de Grand Yoff, Dakar
  - El Hadj-Ibrahima Niass, Kaolack
- National Cardiothoracic center / Shab Teaching Hospital, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marijon E, Ou P, Celermajer DS, Ferreira B, Mocumbi AO, Jani D, Paquet C, Jacob S, Sidi D, Jouven X. Prevalence of rheumatic heart disease detected by echocardiographic screening. N Engl J Med. 2007 Aug 2;357(5):470-6. doi: 10.1056/NEJMoa065085. PMID 17671255
- [Background] Marijon E, Celermajer DS, Tafflet M, El-Haou S, Jani DN, Ferreira B, Mocumbi AO, Paquet C, Sidi D, Jouven X. Rheumatic heart disease screening by echocardiography: the inadequacy of World Health Organization criteria for optimizing the diagnosis of subclinical disease. Circulation. 2009 Aug 25;120(8):663-8. doi: 10.1161/CIRCULATIONAHA.109.849190. Epub 2009 Aug 10. PMID 19667239
- [Background] Marijon E, Mirabel M, Celermajer DS, Jouven X. Rheumatic heart disease. Lancet. 2012 Mar 10;379(9819):953-964. doi: 10.1016/S0140-6736(11)61171-9. PMID 22405798
- [Background] Ranque B, Menet A, Diop IB, Thiam MM, Diallo D, Diop S, Diagne I, Sanogo I, Kingue S, Chelo D, Wamba G, Diarra M, Anzouan JB, N'Guetta R, Diakite CO, Traore Y, Legueun G, Deme-Ly I, Belinga S, Boidy K, Kamara I, Tharaux PL, Jouven X. Early renal damage in patients with sickle cell disease in sub-Saharan Africa: a multinational, prospective, cross-sectional study. Lancet Haematol. 2014 Nov;1(2):e64-73. doi: 10.1016/S2352-3026(14)00007-6. Epub 2014 Oct 28. PMID 27030156
- [Background] Marijon E, Ou P, Celermajer DS, Ferreira B, Mocumbi AO, Sidi D, Jouven X. Echocardiographic screening for rheumatic heart disease. Bull World Health Organ. 2008 Feb;86(2):84. doi: 10.2471/blt.07.046680. No abstract available. PMID 18297157
- [Background] Yusuf S, Rangarajan S, Teo K, Islam S, Li W, Liu L, Bo J, Lou Q, Lu F, Liu T, Yu L, Zhang S, Mony P, Swaminathan S, Mohan V, Gupta R, Kumar R, Vijayakumar K, Lear S, Anand S, Wielgosz A, Diaz R, Avezum A, Lopez-Jaramillo P, Lanas F, Yusoff K, Ismail N, Iqbal R, Rahman O, Rosengren A, Yusufali A, Kelishadi R, Kruger A, Puoane T, Szuba A, Chifamba J, Oguz A, McQueen M, McKee M, Dagenais G; PURE Investigators. Cardiovascular risk and events in 17 low-, middle-, and high-income countries. N Engl J Med. 2014 Aug 28;371(9):818-27. doi: 10.1056/NEJMoa1311890. PMID 25162888